CLINICAL TRIAL: NCT03105960
Title: Evaluation of Garlic With Lime Juice and Chlorhexidine Mouthwash on Gingival Bleeding in Group of Egyptian Children: A Randomized Clinical Trial
Brief Title: Garlic With Lime Juice and Chlorhexidine Mouthwash
Acronym: mouthwash
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, manal sayed abdel latief, oral and dental medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 151087; 151087 (Registry Identifier: manal sayed)
Record Dates: First submitted 2017-03-21; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Gingival Bleeding
MeSH Terms: conditions — Gingival Hemorrhage | interventions — Chlorhexidine

STUDY DESIGN:
Intervention Model Description: A Randomized Clinical Trial parallel
Who Masked: Participant, Investigator
Masking Description: This was a double-blind study as the investigator was unaware about the sampling of the groups and study subjects were unaware about the mouthwash they were using
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- garlic with lime juice mouthwash (Experimental): garlic with lime juice mouthwash is herbal antimicrobial .children were instructed to rinse for 14 days, twice daily, ,10 ml (undiluted) for 30 second and then expectorate .
  To prepare garlic with lime mouth rinse, 100 g of fresh, washed garlic cloves was macerated in a sterile, ceramic mortar and water was added to obtain a homogenate which was then filtered off with a sterile muslin cloth. the final concentration of the solution was determined to be 1 g/100 ml. About 100 ml of lime juice was extracted from fresh lemons using a juice extractor and added to the garlic extract.
  Interventions: Drug: garlic with lime mouth wash
- chlorhexidine mouthwash (Active Comparator): chlorhexidine is antimicrobial, antiplaque mouthwash 10 ml (undiluted) for 30 second twice daily and then expectorate for 14 days. it is commercial mouthwash
  .
  Interventions: Drug: chlorhexidine

INTERVENTIONS:
Drug: garlic with lime mouth wash — garlic with lime juice is herbal antimicrobial 10 ml (undiluted) for 30s and then expectorate for 14 days.o prepare garlic with lime mouth rinse, 100 g of fresh, washed garlic cloves was macerated in a sterile, ceramic mortar and water was added to obtain a homogenate which was then filtered off with a sterile muslin cloth. the final concentration of the solution was determined to be 1 g/100 ml. About 100 ml of lime juice was extracted from fresh lemons using a juice extractor and added to the garlic extract.
  Other Names: herbal mouthwash
  Arms: garlic with lime juice mouthwash
Drug: chlorhexidine — hlorhexidine is antimicrobial, antiplaque mouthwash 10 ml (undiluted) for 30 second twice daily and then expectorate for 14 days.
  Other Names: antimicrobial mouthwash
  Arms: chlorhexidine mouthwash

SUMMARY:
the study about herbal mouthwash. it is clinical trial .the investigator will compare between chlorhexidine mouthwash and garlic with lime juice mouthwash.and their effect on gingival bleeding and plaque and salivary bacteria.

DETAILED DESCRIPTION:
the study about herbal mouth wash. it is clinical trial .the investigator will compare between chlorhexidine mouthwash and garlic with lime juice mouthwash.and show their effect on gingival bleeding and strepococcus bacteria present in saliva and plaque.

1. Preparation of garlic with lime juice will occur under aseptic condition.and give it to the first group.

   provide chlorhexidine to the second group.
2. Collection of plaque and saliva samples will be obtained from children who fulfilled the inclusion criteria.
3. Asses gingival condition by asking patient.
4. Subjects will be instructed to rinse for 14 days, twice daily.
5. Morning after breakfast and night before going to bed.
6. With 10 ml (undiluted) of the assigned mouthwash for 30 s and then expectorate the rinse.
7. Again after 14 days, the saliva and plaque samples will be taken and inoculated on blood agar plates to determine the colony count and the gingival index by loe and illness will be assessed.

ELIGIBILITY:
Inclusion criteria:

1. Children aged between 9 and 12 years.
2. Children are having normal occlusion (no crowding), non-compromised oral health (brushed their teeth once-daily) using toothbrush and non-fluoridated toothpaste. And practicing no other oral hygiene measures.
3. Medically free history.
4. Absence of orthodontic appliances.

Exclusion criteria:

1. History of current or recent (at least for the past 1 month) antibiotic usage or other medications.
2. Presence of Abscess, draining sinus, cellulitis, or other conditions requiring emergency dental treatment.
3. not willing to comply with the study.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Egyptian children
Enrollment: 36 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2017-06-01 (Estimated); Study Completion 2017-06-01 (Estimated)

PRIMARY OUTCOMES:
gingival bleading | 15 day
  bleeding of gingiva asses by yes or no

SECONDARY OUTCOMES:
Streptococcal count in saliva and plaque | 15 day
  Streptococcal count in saliva and plaque

CONTACTS AND LOCATIONS:
Overall Officials: sherif B eltweel, Ass.prof, Study Director — Cairo univaesity
Locations (1):
- Manal Sayed Abdel Latief, Helwan, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
it will be available when it finish

REFERENCES:
- [Background] Tulsani SG, Chikkanarasaiah N, Siddaiah SB, Krishnamurthy NH. The effect of Propolis and Xylitol chewing gums on salivary Streptococcus mutans count: a clinical trial. Indian J Dent Res. 2014 Nov-Dec;25(6):737-41. doi: 10.4103/0970-9290.152182. PMID 25728105
- See also: Description related info — http://doi.org/10.4103/0970-9290.152182